CLINICAL TRIAL: NCT04228276
Title: Treating Stimulant Addiction With Repetitive Transcranial Magnetic Stimulation
Acronym: VA-StARTS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic adversely affected recruitment.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3314-P; 54458 (Other: Stanford University)
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Stimulant Use Disorder; Substance-related Disorders
Keywords: Magnetic resonance imaging; Transcranial magnetic stimulation; Dopamine; Reward processing
MeSH Terms: conditions — Substance-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups to receive active or sham rTMS.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Experimental): Receive active rTMS
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Sham rTMS (Sham Comparator): Receive sham rTMS
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — rTMS is a non-invasive procedure in which administering a transient magnetic field induces electrical currents in specific, targeted brain regions. The intervention (active and sham) will be administered in 8 sessions across 2 weeks. The brain region targeted is the dorsolateral prefrontal cortex.

SUMMARY:
The purpose of this study is to establish a new treatment (repetitive transcranial stimulation (rTMS)) for Veterans with stimulant use disorder (SUD). Despite the large public health burden imposed by SUD, there is currently no FDA-approved or widely recognized effective somatic treatment. rTMS may be a promising treatment option for SUD. In this study, we will demonstrate the feasibility of applying rTMS to Veterans with SUD, examine the efficacy of rTMS in the treatment of SUD, and explore biomarkers that may guide patient selection for rTMS treatment and predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Structured Clinical Interview for DSM Disorders (SCID) confirmed diagnosis of SUD, severe
* Last use of stimulants >1 and <6 weeks
* Stable medication regimen (no change in dose or agents between 2 weeks prior to the start of and throughout the treatment phase of the study)
* Stable social environment and housing to enable regular attendance at clinic visits.
* Ability to undergo cognitive testing, functional magnetic resonance imaging (fMRI) scans, and rTMS (no contraindications)
* Intelligence Quotient (IQ) > 80
* Stable medical health
* Veteran at Palo Alto VA's Addiction Treatment Services

Exclusion Criteria:

* Pregnant or lactating female
* History of prior adverse reaction to TMS
* On medications thought to significantly lower seizure threshold, e.g.:

  * clozapine
  * chlorpromazine
  * clomipramine
  * bupropion > 400 mg/day
* Use of direct dopaminergic antagonists or agonists
* History of seizures or conditions known to substantially increase risk for seizures
* Implants or medical devices incompatible with TMS
* Acute or unstable chronic medical illness that would affect participation or compliance with study procedures, e.g. unstable angina
* Unstable psychiatric symptoms that precludes consistent participation in the study, e.g.:

  * active current suicidal intent or plan
  * severe psychosis
* Inability to undergo fMRI scan, e.g. claustrophobia, presence of ferromagnetic objects in subject's body
* Other substance use disorder not in sustained remission
* Chronic or recurring Axis I psychiatric condition preceding SUD other than PTSD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong H. Yoon, MD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 people did not enter intervention phase. Defining drop out as those who started the intervention and dropped out before completing intervention & outcome measures.
Groups:
- Active rTMS: Receive active rTMS
  Repetitive transcranial magnetic stimulation (rTMS): rTMS is a non-invasive procedure which administers a transient magnetic field inducing electrical currents in specific, targeted brain regions. The intervention was administered in 8 sessions across 2 weeks. The brain region targeted is the dorsolateral prefrontal cortex.
- Sham rTMS: All subjects underwent the same procedure as the active rTMS group except that the inactive side of the coil was placed on the subject's scalp. The experience receiving sham rTMS was identical except that no electrical current was administered.
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 9 | 13
Completed | 7 (Primary completion: 04/30/2024) | 11
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Data is only available for participants who completed intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Continuous [Mean (Standard Deviation); unit: Year] | 40.4 (11.3) | 45.0 (16.9) | 43.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Relapsed
Description: Rate of stimulant use relapse compared between active vs. sham rTMS groups
Time Frame: 3 months after last rTMS treatment
Measure: Count of Participants; unit: Participants
Groups:
- Sham TMS: All subjects underwent the same procedure as the active rTMS group except that the inactive side of the coil was placed on the subject's scalp. The experience receiving sham rTMS was identical except that no electrical current was administered.
Arm/Group | Active rTMS | Sham TMS
Number analyzed (Participants) | 7 | 11
Participants | 4 | 8

2. Secondary Outcome: Reward Circuit Function and Signaling
Description: Before and after treatment, participants underwent functional magnetic resonance imaging (fMRI) imaging while completing the Monetary Incentive Delay Task, a validated probe of reward processing circuit function and dysfunction. Signaling in the substantia nigra measured in an individual-subject, "native space" region of interest approach as a marker of dopaminergic reward processing function, as well as in voxel-wise, whole-brain exploratory analyses. Changes in reward function and signaling compared between active vs. sham rTMS groups
Time Frame: Within 1 week before and after rTMS treatment
Population: Unable to conduct this portion of study due to COVID-19 pandemic related logistical challenges. Data will never be collected in the future.
Arm/Group | Active rTMS | Sham TMS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/11
Other Adverse Events (participants affected / at risk) | 0/7 | 0/11

LIMITATIONS AND CAVEATS:
COVID-19 pandemic adversely affected recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-04-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04228276/Prot_001.pdf
  • Statistical Analysis Plan (2025-04-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04228276/SAP_002.pdf
  • Informed Consent Form (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT04228276/ICF_000.pdf